CLINICAL TRIAL: NCT03527355
Title: A Phase II, Randomized, Dose-scheduling, Observer-Blinded Study to Assess the Safety, Reactogenicity and Immunogenicity of Vi-DT Conjugate Vaccine in 6-23-Month Old Healthy Filipino Infants and Toddlers
Brief Title: Safety, Reactogenicity and Immunogenicity of Vi-DT;Typhoid Conjugate Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: SK Bioscience Co., Ltd. (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI T002
Record Dates: First submitted 2018-02-12; First posted 2018-05-17 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2020-04

CONDITIONS: Typhoid
Keywords: Typhoid; Vi-DT; Conjugate vaccine; First in human; New vaccine
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Intervention Model Description: Participants age 6-23 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Single dose) (Experimental): One dose of Vi-DT (Typhoid conjugate vaccine) 25 µg 0.5 mL is administrated intramuscularly at first dost (Day 0).
  One dose of FluQuadri™ 0.25mL is administrated intramuscularly at second dose (Week 24).
  One booster dose of Vi-DT 0.5 mL is administrated 2 years apart (Week 96). MMR for age group at 9-12 months.
  Interventions: Biological: Vi-DT; Biological: FluQuadri™
- B (Two dose) (Active Comparator): Two doses of Vi-DT (Typhoid conjugate vaccine) 25 µg 0.5 mL is administrated intramuscularly 6 months apart (Day 0 and Day 168 (Week 24)).
  MMR for age group at 9-12 months.
  Interventions: Biological: Vi-DT
- C (Placebo/Comparator) (Placebo Comparator): One dose of Placebo (0.9% sodium chloride isotonic solution) 0.5 mL is administrated intramuscularly at first dost (Day 0).
  One dose of FluQuadri™ 0.25mL is administrated intramuscularly at second dose (Day 168; Week 24).
  MMR for age group at 9-12 months.
  Interventions: Biological: FluQuadri™; Other: 0.9% sodium chloride isotonic solution

INTERVENTIONS:
Biological: Vi-DT — Manufacturer: SK Bioscience Co., Ltd. Ingredient: Purified Vi-polysaccharide conjugated to diphtheria toxoid Dose: 0.5 mL/Vial
  Other Names: Vi-DT typhoid conjugate vaccine
  Arms: A (Single dose); B (Two dose)
Biological: FluQuadri™ — Manufacturer: Sanofi Pasteur Dose: 0.25 ml
  *Participants who have not been vaccinated for flu before, will receive a second dose of flu-vaccine after unblinding.
  Arms: A (Single dose); C (Placebo/Comparator)
Other: 0.9% sodium chloride isotonic solution — Manufacture: Euro-Med Inc. Dose: 0.5 mL
  Arms: C (Placebo/Comparator)

SUMMARY:
This is a randomized, observer-blinded Phase 2 study in healthy infants and toddlers 6-23 months of age at the time of the first vaccine dose.

The purpose of this study is to assess the safety and immunogenicity of the Vi-DT vaccine in age group 6-23months of age.

The Vi-DT vaccine is administered at 25 µg either as a single dose, or two doses given 6 months apart.

DETAILED DESCRIPTION:
This study is carried out in healthy children aged 6 to 23 months at a single site. A total of 285 participants are enrolled, 114, 114 and 57 participants are randomized to either the single dose, two-dose Vi-DT regimens or placebo/comparator group, respectively within age strata. Three age strata is 6 to less than 9 months, 9 to 12 months and 13 to 23 months. The investigators allow the 9-12 months old children to receive Measles-Mumps-Rubella (MMR) vaccine concomitantly with Vi-DT vaccine and descriptive analysis of immune response to MMR only and to MMR and Vi-DT vaccines are performed to assess the possible immunological interference with MMR vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants and children 6-23 months of age at enrollment as determined by medical history, physical examination and clinical judgment of the investigator
* Birth weight ≥ 2500 g
* ≥ 37 weeks of pregnancy or judge to be full-term by the midwife or birth attendant
* Parents aged 18 years and above and legal guardians aged 21 years and above as per the legal authorization in the Philippines, who have voluntarily given informed consent
* Parents/ legal guardians willing to follow the study procedures of the study and available for the entire duration of the study

Exclusion Criteria:

* Child with a congenital abnormality
* Subject with abnormal routine biological values at screening
* Subject concomitantly enrolled or scheduled to be enrolled in another trial
* Acute illness, in particular infectious disease or fever (axillary temperature ≥37.5°C), within three days prior to enrolment and vaccination
* Known history of immune function disorders including immunodeficiency diseases, or chronic use of systemic steroids (>20 mg/day prednisone equivalent for periods exceeding 10 days), cytotoxic or other immunosuppressive drugs
* Child with a previously ascertained or suspected disease caused by S. typhi
* Child who have had household contact with/and or intimate exposure to an individual with laboratory-confirmed S. typhi
* Known history or allergy to vaccines or other medications
* Know history of allergy to eggs, chicken protein, neomycin and formaldehyde
* History of uncontrolled coagulopathy or blood disorders
* Mother has known HIV infection or other immune function disorders
* Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the subject and interfere with the assessment of the study objectives
* Child whose parents or legal guardian planning to move from the study area before the end of study period

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-07-28 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Safety endpoints: solicited and unsolicited adverse events and serious adverse events | Solicited AE: during 7 days after each vaccination. Unsolicited AE: after the first vaccination until 4 weeks after the second vaccination. SAE will be captured after the first vaccination up to week 100 for Group A, week 96 for Group B, week 36 Group C
  * Frequency (percentage) of solicited local reactions at the injection site: Pain, tenderness, erythema/redness, swelling/induration and pruritus local
  * Frequency (percentage) of solicited systemic reactions: Fever, lethargy, irritability, vomiting, diarrhea, drowsiness, loss of appetite, persistent crying, rash and nasopharyngitis
  * Frequency (percentage) of unsolicited adverse events
  * Frequency (percentage) of serious adverse events

SECONDARY OUTCOMES:
Immunogenicity Endpoints | At week 28, 4 weeks after the second vaccination
  Seroconversion rate of anti-Vi IgG by Geometric Mean Titers (GMT) will be measured 4 weeks after the second vaccination using an in-house ELISA assay using standardized reagents and reference serum. The level of the specific anti-Vi IgG in ELISA units for each serum sample is determined by comparison to a reference serum. The number of anti-Vi IgG positive sera will be used to calculate the seroconversion rates.

OTHER OUTCOMES:
Exploratory Endpoints | At week 4, 4 week after MMR vaccination
  Seroconversion rates of Measles, Mumps and Rubella will be determined 4 week after MMR vaccination. Serum titers will be measured by routinely used commercially available ELISA kits. Kit-specific threshold of positivity will be used to determine specific seroconversion rates.
Exploratory Endpoints | At week 28, 4 weeks after the second vaccination and at week 96 after the booster dose in selected group.
  Serum bactericidal titers will be determined using in-house functional assay assessing the number of survived S. Typhi Ty2 strain colony on Luria-Bertani plate. Serum bactericidal titer is defined as the highest dilution of serum that gives 50% of inhibition of colony formation of S. Typhi.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario Capeding, MD, Principal Investigator — Research Institute for Tropical Medicine, Metro Manila, Philippines
Locations (1):
- Research Institute for Tropical Medicine(RITM), Alabang, Muntinlupa City, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capeding MR, Sil A, Tadesse BT, Saluja T, Teshome S, Alberto E, Kim DR, Park EL, Park JY, Yang JS, Chinaworapong S, Park J, Jo SK, Chon Y, Yang SY, Ryu JH, Cheong I, Shim KY, Lee Y, Kim H, Lynch JA, Kim JH, Excler JL, Wartel TA, Sahastrabuddhe S. Safety and immunogenicity of Vi-DT conjugate vaccine among 6-23-month-old children: Phase II, randomized, dose-scheduling, observer-blind Study. EClinicalMedicine. 2020 Sep 9;27:100540. doi: 10.1016/j.eclinm.2020.100540. eCollection 2020 Oct. PMID 33150320
- [Derived] Capeding MR, Alberto E, Sil A, Saluja T, Teshome S, Kim DR, Park JY, Yang JS, Chinaworapong S, Park J, Jo SK, Chon Y, Yang SY, Ham DS, Ryu JH, Lynch J, Kim JH, Kim H, Excler JL, Wartel TA, Sahastrabuddhe S. Immunogenicity, safety and reactogenicity of a Phase II trial of Vi-DT typhoid conjugate vaccine in healthy Filipino infants and toddlers: A preliminary report. Vaccine. 2020 Jun 9;38(28):4476-4483. doi: 10.1016/j.vaccine.2019.09.074. Epub 2019 Oct 1. PMID 31585725
- See also: A preliminary report — https://doi.org/10.1016/j.vaccine.2019.09.074